CLINICAL TRIAL: NCT02675673
Title: A Randomized Comparison of Enteral Feeding for Head and Neck (HNC) Cancer Patients
Brief Title: Feeding Tube in Cancer Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Logistical issues
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UHN REB 08-0393-CE
Record Dates: First submitted 2013-06-11; First posted 2016-02-05 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: Enteral Feeding for Head and Neck Cancer Patients
Keywords: Enteral Feeding; G-Tube; GJ Tube
MeSH Terms: interventions — Gastrostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GJ-Tube arm (Active Comparator): Patients randomized to his arm would usually have a small tube is inserted through the nose into the stomach first, so that air can be used to fill the stomach to make it visible on X-ray. A fine needle is then used to inject freezing medicine (local anesthetic) into the skin of the abdomen. Using an x-ray machine for guidance, a puncture is made into the stomach through the frozen skin. The feeding tube is placed through this puncture into the stomach and the tube tip is placed in the small bowel. Once the GJ-tube has been inserted, the tube in the nose is removed.
  Interventions: Procedure: GJ-Tube
- G-Tube arm (Active Comparator): Patients who are randomized to this arm will usually have a small tube is inserted through the nose into the stomach first, so that air can be used to fill the stomach to make it visible on X-ray. A fine needle is then used to inject freezing medicine (local anesthetic) into the skin of the abdomen. Using an x-ray machine for guidance, a puncture is made through the frozen skin. A small guiding tube or catheter is placed through this puncture into the stomach, and is advanced up the esophagus and out of the mouth. The feeding tube is then pulled into the mouth, down the esophagus, and positioned through the abdomen with its inside tip in the stomach.
  Interventions: Procedure: G-Tube

INTERVENTIONS:
Procedure: GJ-Tube — Insertion of a GJ tube either prior to the start of radiotherapy or within the first 2 weeks after the first dosage.
  Arms: GJ-Tube arm
Procedure: G-Tube — Insertion of a G-tube either prior to the start of radiotherapy or within the first 2 weeks after the first dosage.
  Arms: G-Tube arm

SUMMARY:
The purpose of this study is to compare the quality of life (QOL) in head and neck patients who are given the GJ tube (which is placed in the bowel) versus those who are given the G-Tube (which is placed in the stomach) for prophylactic feeding. The standard of care for patients at Princess Margaret Hospital (PMH) is using GJ tubes. Patients who agree to be in the study will be randomized to either the GJ-Tube or the G-Tube arm. Patients randomized to the G-tube will receive prophylactic intravenous and oral antibiotics prior to insertion of the G-tube. Antibiotics will be given for a total of 1 week. A few hours following tube insertion (on return to PMH ward), patients will complete a single item, visual analogue pain scale (VAS). Patients will remain in hospital for a minimum of 24 hours and until the patient and/or family is able to care for the Enteric Feeding(EF) device at home. Patients randomized to the GJ-Tube may receive i.v medication during the procedure. All Patients will be asked to fill out several questionnaires at different time- points of the study. All Patients will have regular assessments to evaluate their overall quality of Life, toxicity, and how they respond to treatment during the study. Patients will also be assessed after they completed study treatment.

DETAILED DESCRIPTION:
Prophylactic enteral feeding tubes are used routinely for nutritional support during intensive radiotherapy or chemoradiotherapy for locally advanced head and neck cancer. Typically, tubes remain in place for up to 3-4 months. Whether small-bore jejunal (GJ) or larger bore gastric (G) tubes are used varies geographically, based on tradition, physician preference and availability of services. Feeding tube placement is arranged either prior to the start of RT, or more commonly within the first 2 weeks of RT, prior to the onset of severe mucositis. Patients are admitted to hospital for 1-3 days to monitor side effects of the procedure, and to allow our dietetic and nursing staff to provide intensive teaching on the use and care of the tube. Feeding tubes are kept in place through the treatment course and removed once patients are able to meet their calorie needs and maintain body weight through oral feeding. On average, feeding tubes are removed approximately 2-3 months after completion of RT; however, approximately 20% of patients may still require enteral feeding at 1 year post-treatment. This study will compare the QOL in patients who use the G tube versus the GJ tube.

ELIGIBILITY:
Inclusion Criteria:

* local regional carcinoma of the oral cavity, pharynx, paranasal sinuses, larynx, cervical esophagus
* patients who will receive potentially curative radiotherapy or chemotherapy
* patients who are recommended for prophylactic enteral feeding

Exclusion Criteria:

* patients who are unable to give consent
* patients who have other concurrent active cancer diagnosis
* patients with established pharyngeal obstruction and/or presence of an EF device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-09; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Quality of Life questionnaire: Enteric Feeding (QOL-EF) | 1 year
  A 20-item specific questionnaire scored using individual items from 1=not at all to 5=very much

SECONDARY OUTCOMES:
Evaluation of post-procedure pain associated with the use of feeding tubes | 1 year
  Visual analog scale
Quality of Life questionnaire: M.D.Anderson Swallowing Inventory (MDADI) | 1 year
  A self-reported utility consisting of 20 discrete 5-level items rated from "strongly agree" to "strongly disagree"
Patient weight loss associated with the use of feeding tubes | 2 years
  weight will be measured at protocol-determined time points
Quality of Life questionnaire: Functional Assessment of Cancer Therapy (FACT-HN) | 1 year
  •Quality of life as measured by Functional Assessment of Cancer Therapy-Head & Neck (FACT-HN) ranking 24 individual items from 0= not at all to 4 = very much
Symptoms associated with the use of feeding tubes (as per CTCAE v4 criteria) | 1 year
  Clinical toxicities will be grade according to Common Terminology Criteria for Adverse Events version 4.03 (CTCAE v4), a well known toxicity grading scale from 0 (asymptomatic) to 5 (death)

CONTACTS AND LOCATIONS:
Overall Officials: Jolie Ringash, MD, Principal Investigator — University Health Network, Princess Margaret Hospital